CLINICAL TRIAL: NCT07336108
Title: RUG-WEAVING PLICATION TECHNIQUE RESULTS IN CYSTOCELE TREATMENT:TWO YEAR FOLLOW-UP
Brief Title: RUG-WEAVING PLICATION IN CYSTOCELE TREATMENT
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Bedir Fındık, DR, Ankara City Hospital Bilkent
Other Study IDs: There is no sponsor.
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:there were data of 29 patients who were operated for cystocele with the Rug Wave techniq: Rug Waiving plication techniqe
  Interventions: Procedure: rug weaving-like plication technique
- Group 2: 31 patients who underwent surgery using conventional colporrhaphy.: anterior vaginal wall repair with theconventional technique in cystosel
  Interventions: Procedure: group 2:conventional technique cystocele treatment

INTERVENTIONS:
Procedure: rug weaving-like plication technique — Rug Waeving plication technique :This technique is a technique that has not been used before.
  Groups: Group 1:there were data of 29 patients who were operated for cystocele with the Rug Wave techniq
Procedure: group 2:conventional technique cystocele treatment — Patients operated on using the conventional anterior colporrhaphy
  Groups: Group 2: 31 patients who underwent surgery using conventional colporrhaphy.

SUMMARY:
In this study was to compare the 2-year results of the Rug Wave plication technique, which it present as a natural tissue repair technique in cystocele, with the conventional technique in terms of both recurrence and patient quality of life satisfaction scales.

DETAILED DESCRIPTION:
The study was planned as a retrospective case-control observational study. It included 60 patients who underwent surgery solely for cystocele or cystocel with other organ prolapse conditions; of them, 29 received the rug-weaving plication technique, a natural tissue repair method implemented for anterior wall defects since 2022, and 31 underwent conventional anterior colporrhaphy.Data were collected in 2 groups. In Group 1, there were data of 29 patients who were operated for cystocele with the Rug Wave technique and Group 2, there were data of 31 patients who were operated with the classical colporrhaphy technique. Data from these patients were recorded at 6 months and 2 years postoperatively. At the 6 months and 2 years postoperative follow-up, it assessed patients' complaints, degree of prolapse (using the simplified Pelvic Organ Prolapse Quantification system), pelvic floor muscle strength (using the Modified Oxford Score) and the anterior vaginal wall thickness in transvaginal ultrasound. In addition, the data of the questionnaire applied to the patients in the 2nd year were also recorded(Pelvic Floor Distress Inventory, Sandvik Severity Index, Overactive bladder, Surgical satisfaction questionnaire, Patient global impression of improvement questionnaire, Pelvic Organ Prolapsed / Urinary Incontinence Sexual Questionnaire, Incontinence Impact Questionnaire).The results of the two groups were compared.Data were entered and analyzed in SPSS program. Mann-Whitney -U test, Independent simple test, Chi-Square test were used in group comparisons. Chi-Square test was used to compare categorical variables; Mann-Whitney U test was used to compare continuous variables that were not normally distributed; Independent Simple test was used to evaluate the significance of the differences between the means of continuous variables between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on using the rug weaving plication technique
* Patients operated on using the conventional anterior colporrhaphy

Exclusion Criteria:Patients who did not undergo cystocele surgery were excluded from the study.

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Women operated on for anterior wall prolapse in POP-Q
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) Postoperative anterior wall POP-Q | 2 years
  The POP-Q staging system, introduced in 1996 and widely accepted as the standard quantitative classification system for pelvic organ prolapse, was utilized in this study. Measurements were conducted with a scaled abeslang while the patient was in the lithotomy position. Evaluation of the anterior compartment involved measuring points Aa and Ba, the apical compartment involved points C and D, and the posterior compartment involved points Ap and Bp. Staging was determined based on the lowest point of prolapse. Stage 0 indicated normal pelvic floor support, Stage 2 indicated a distance between -1 and 1 from the hymen, and Stage 4 indicated total uterine prolapse (prosidentia). Stages 1,2 and 3 indicated intermediary levels of prolapse severity, counting for grades between Stage 0 and 4. Figure -1 schematically shows the POP-Q staging system .

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to patient privacy

REFERENCES:
- [Background] Findik RB, Doganay M, Aksakal OS, Coskun ZY, Karakaya J. A novel suturing technique for natural tissue repair in cystocele treatment. BMC Womens Health. 2024 Aug 29;24(1):474. doi: 10.1186/s12905-024-03317-3. PMID 39210362